CLINICAL TRIAL: NCT06984016
Title: Photogrammetry Analysis in the Assessment of Work-related Musculoskeletal Disorders Risk Among Physical Therapists
Acronym: WRMD
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, alaa mohamed ibrahim hashem, principle investigator : alaa mohamed ibrahim, Cairo University
Other Study IDs: 012/005703
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Musculoskeletal Disorder
Keywords: Photogrammetry Analysis; physical therapist; Musculoskeletal Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Work-related Musculoskeletal Disorders Risk Among Physical Therapists: The study will be carried out on 217 of Egyptian physical therapists . They will be randomly selected from Al Kasr Elaini Hospital and at the outpatient clinics of the Faculty of Physical Therapy at Cairo and Badr University.
  Interventions: Other: Work-related Musculoskeletal Disorders Risk Among Physical Therapists

INTERVENTIONS:
Other: Work-related Musculoskeletal Disorders Risk Among Physical Therapists — 217 Males and females Egyptian physical therapists at will be included in the study.

SUMMARY:
this study will be conducted to investigate the risk of work-related musculoskeletal disorders due to the postural load among physical therapists

DETAILED DESCRIPTION:
Musculoskeletal disorders (MSDs)refer to an array of signs and symptoms involving various areas of the musculoskeletal system. The clinical manifestations of MSDs include pain, swelling/redness, stiffness, and weakness or loss of function. Such manifestations affect the muscles, joints, tendons, nerves, and supporting structures in various body parts. Work-related musculoskeletal disorders (WMSDs) have a high significant occupation problem worldwide. One-third of all injuries in a day occurs due to occupational hazards are WMSDs reports The Bureau of Labor Statistics.Previous works have shown that parameters such as the environment , the level of experience , the country of origin ,the institution in which the professional evolves had an influence on the level of risk of WMSD prevalence. Many studies have addressed the issue of WMSD in PPTs. The prevalence of MSDs by body area is the most commonly used analysis . The results showed that the areas most at risk for MSDs are the neck, lower back and upper extremities. However, the studies reported different results. Indeed, the prevalence vary between 5.3 % and 61 % , between 14.3 % and 62 % and 8 % and 83 % respectively for the neck, low back and thumb. These differences in prevalence have also been observed in other areas such as the shoulder or lower extremity . Studies have focused on risk factors responsible for the occurrence of MSD or which reinforce the associated symptoms. two hundreds supjects will be conducted to this study

ELIGIBILITY:
Inclusion Criteria:

* Males and females Egyptian physical therapists at Al Kasr Elaini Hospital and at the outpatient clinics of the Faculty of Physical Therapy, Cairo University, and Badr university, will be included in the study.
* Age ranges from 21-30 years old of physical therapists and their BMI is between 18 and 24.9.
* 4 hours of work daily at least
* No working experience to 2 years of experience only

Exclusion Criteria:

* Congenital musculoskeletal disorders
* Fractures
* Previous musculoskeletal surgery
* Cardiovascular disease
* Pulmonary disease
* Diabetes
* Neurological disease

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 217 Males and females Egyptian physical therapists at Al Kasr Elaini Hospital and at the outpatient clinics of the Faculty of Physical Therapy, Cairo University, and Badr university, will be included in the study.
Sampling Method: Probability Sample
Enrollment: 217 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
range of motion | up to thirty minutes
  kinovea soft wear will be used to measure joints range of motions.this will be applied through Capturing videos by iPhone 11 from lateral view for kinovea analysis the angles degrees of sagittal plane motion (for shoulder , elbow, wrist, neck and trunk joints ) and from anterior view to determined the presence of frontal plane motion (in shoulder, elbow, wrist, neck and trunk joints)
postural load | up to thirty four weeks
  • The rapid upper limb assessment (RULA) will be used to assess the postural load and to know if physical therapy interns are exposed to MSD risk factors during the performance of their work